

# TC KÜTAHYA HEALTH SCIENCES UNIVERSITY RECTORATE NON-INTERVENTIONAL CLINICAL RESEARCH ETHICS COMMITTEE APPLICATION FORM

| 1. 1. APPLICATION PETITION ( signed ) | $\boxtimes$ |
|---|---|
| 2. 2. APPLICATION CONTENT FORM | $\boxtimes$ |
| 3. APPLICATION FORM (fully filled) | $\boxtimes$ |
| 4. COMMITMENT ( Must be signed by the entire research team) | $\boxtimes$ |
| 4. RESEARCH BUDGET (The budget source has been specified, including all the expenditures to be | $\boxtimes$ |
| made-<br>(included in the application form ) | |
| 5. CVs (belonging to all researchers participating in the study) | |
| 6. INFORMED VOLUNTEER CONSENT FORM (If it is planned to include volunteers under the age of 18, a child consent form and a parent/guardian consent form should also be prepared) | |
| 7. MATERIAL PURCHASE CONSENT FORM (if necessary) | |
| 8. USED SURVEY ETC. FORMS (All forms must be attached) | $\boxtimes$ |
| 9. CERTIFICATE OF APPROVAL OF THE HEADS OF THE RELEVANT DEPARTMENT / LABORATORY RESPONSIBILITIES | |
| 10. INSTITUTIONAL PERMISSION CERTIFICATE (If the approval of the head of the department, the approval of the other department heads + the approval of the Chief Physician) | |
| ( If the institution is different, approval of the department head + approval of the relevant institution (such as MEB)) | |
| 11. APPROVAL LETTER THAT YOU ARE A STUDENT OF THE RELATED INSTITUTE (if the research is a thesis and the researcher is an institute student) | |
| 12. 3 PUBLICATIONS RELATED TO THE RESEARCH (Article published in full text) | $\boxtimes$ |
| 13. DATA SECURITY AGREEMENT (For research where necessary) | |
| 14. COMMITMENT TO IKU, İLU AND HELSINKI DECLARATION (Signed by all investigators participating in the study ) | |
| 15 . Delivery of the application file to the Ethics Committee secretariat | $\boxtimes$ |

#### Tick the relevant boxes with a cross.

Studies with missing application forms will not be evaluated. I undertake that I have submitted all documents in full.

Name of the Study: Evaluation of the Effect of Watching Surgery Videos on Social Media on Anxiety Before

**Impacted Wisdom Tooth Extraction** 

Principal Researcher: Dr. Lecturer Berkan Altay

**Signature and Date:** 



# TR KÜTAHYA HEALTH SCIENCES UNIVERSITY RECTORATE

# NON-INTERVENTIONAL CLINICAL TRIALS TO THE ETHICS COMMITTEE

I would like to submit your information and the need for your committee to review our research titled '
Evaluation of the Effect of Watching Surgery Videos on Social Media on Anxiety Before Impacted
Wisdom Tooth Extraction'.

Responsible Researcher
Dr. Lecturer Berkan Altay
Date and Signature

### TR KÜTAHYA HEALTH SCIENCES UNIVERSITY RECTORATE NON-INTERVENTIONAL CLINICAL TRIALS ETHICS COMMITTEE APPLICATION CONTENT FORM

Name of the Researcher : Dr. Lecturer Berkan Altay
Name of the Research : Evaluation of the Effect of Watching Surgery Videos on Social Media on Anxiety Before Impacted Wisdom Tooth Extraction

| Scope | | |
|---|---|---|
| observational studies | Descriptive | |
| | cross-sectional | |
| | case-control | |
| | Prospective cohort | + |
| | retrospective cohort | |
| | Other (specify) | |
| methodological | + | |
| Survey studies | + | |
| Retrospective archive scans such as file and image recordings | | |
| with biochemistry, microbiology, pathology, and radiology collection materials such as blood, urine, tissue, radiological image or materials obtained during routine examination, examination, analysis and treatment procedures | | |
| Cell or tissue culture studies | | |
| Studies to be carried out with genetic material that are outside of gene therapy clinical studies and for identification purposes, | | |
| Research on body physiology such as exercise | | |
| Studies based on anthropometric measurements | | |
| All research that does not require the direct intervention of<br>a physician, such as research on the evaluation of living<br>habits. | + | |
| New scale development | | |

# APPLICATION FORM

# A. TITLE OF THE SURVEY

| <b>A.1</b> | SCIENTIFIC NAME OF THE RESEARCH Evaluation of the effect of watching surgery videos on social media on anxiety before impacted wisdom tooth extraction | |
|---|---|---|
| A.2 | PUBLIC NAME OF THE RESEARCH It was aimed to evaluate the effect of watching surgery videos on social media on patients' anxiet before impacted wisdom tooth extractions. | ty |
| A.3 | FEATURE OF THE RESEARCH | |
| A.3.1 | master's thesis | |
| A.3.2 | PhD thesis | |
| A.3.3 | Master thesis | |
| A.3.4 | Individual research project | $\boxtimes$ |
| A.3.5 | If other, please specify. | |

### **B. RESEARCH TEAM**

| B.1 | RESP | ONSIBLE RESEARCHER | | |
|---|---|---|---|---|
| B.1.1 | Title, | Name Surname: Dr. Lecturer Berkan Altay | | |
| B.1.2 | | f Specialization and Workplace: <b>Oral, Dental an</b> esity <b>Faculty of Dentistry</b> | d Max | xillofacial Surgery- Kütahya Health Sciences |
| | Role in | the Project: | | |
| | | hypothesis development | | Planning |
| B.1.3 | | Data acquisition | $\boxtimes$ | Data analysis and interpretation |
| | | report writing | | Other, specify |
| | | Critical evaluation of the article report | | |
| B.1.4 | E-mail | l address and GSM No: berkan.altay@ksbu.edu | <u>ı.tr</u> 053 | 356557441 |
| B.2 | ASSIS | STANT RESEARCHER | | |
| B.2.1 | Title, | Name Surname: Dr. Lecturer Mohammad Na | ıbi Ba | siry |
| B.2.2 | | of Specialization and Workplace: Oral, Denta<br>es University Faculty of Dentistry | l and | Maxillofacial Surgery- Kütahya Health |

| | Role in | n the Project: | | |
|---|---|---|---|---|
| | | hypothesis development | | Planning |
| B.2.3 | | Data acquisition | | Data analysis and interpretation |
| | $\boxtimes$ | report writing | | Other, specify |
| | $\boxtimes$ | Critical evaluation of the article report | | |
| <b>B.2.4</b> | E-mail | address and GSM No: mohammednabi.basiry | <u>@ksbu</u> | <u>ı.edu.tr</u> 05079321384 |
| B.3 | ASSIS | STANT RESEARCHER | | |
| B.3.1 | Title, | Name Surname: <b>Dt . Seyma Kale</b> | | |
| B.3.2 | Field o | of Specialization and Workplace: <b>Oral, Denta</b><br>es University Faculty of Dentistry | al and | Maxillofacial Surgery- Kütahya Health |
| | in the | Project : | | |
| | | hypothesis development | | Planning |
| B.3.3 | | Data acquisition | | Data analysis and interpretation |
| | | report writing | | Other, specify |
| | | Critical evaluation of the article report | | |
| B.3.4 | E-mail | address and GSM No: <a href="mailto:seyma.kale@ksbu.edu">.seyma.kale@ksbu.edu</a> | <u>.tr</u> 055 | 333618111 |
| <b>B.4</b> | ADVI | SOR | | |
| B.4.1 | Title, | Name Surname: | | |
| B.4.2 | Area o | of Expertise and Workplace: | | |
| | Topics | Discussed: | | |
| | | Scientific | | Planning |
| B.4.3 | | Translation | | Statistics |
| | | Technical | | Other, specify |
| | | finance | | |
| B.4.4 | E-mail | address and GSM No: | | |

# C. RESEARCH INFORMATION

| | GENERAL INFORMATION |
|---|---|
| C.1 | Surgical extraction of impacted wisdom teeth creates a high level of anxiety on patients. Anxiety in patients can affect the difficulty of tooth extraction, prolong the duration of surgery and increase post-operative pain. With the increasing internet usage in recent years; patients can access different information about surgical procedures by watching videos on various social media platforms in an uncontrolled manner. In the literature, the effects of impacted tooth extraction videos, which are watched by physicians before the operation, on anxiety have been examined. However, studies on |

the evaluation of the effect of the surgery videos watched by the patients before the surgery on their own desires on anxiety and pain perception have been limited.

#### PURPOSE OF THE RESEARCH

**Study Purpose:** It was aimed to evaluate the effects of watching videos with images of the surgery on social media before the impacted tooth extraction operation on anxiety.

#### **METHODS and MATERIALS**

The study was given to KSBU Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery; It will be applied to patients who are referred from Oral, Dental and Maxillofacial Radiology and who want to participate in the study. In our study, the Situational-Trait Anxiety Inventory will be used to assess anxiety. Patients who are referred to our clinic from Oral, Dental and Maxillofacial Radiology and who have impacted wisdom teeth will be evaluated in terms of extraction indication. Patients with an indication for extraction will be asked to score the sentences in the Situational and Trait Anxiety Inventory in that session in order to make an appointment for surgery (Survey 1). Patients will be informed about impacted tooth extraction as routinely practiced. Within the scope of this study, no information about the extraction will be given in the Oral, Dental and Maxillofacial Radiology clinic, standard information will be given to the patients in our clinic and the surgery appointment will be given one week later. On the day of tooth extraction, patients will be asked whether they watched a video about impacted tooth extraction from any social media platform. The patients who watch the video will be assigned to the study group, and the patients who do not watch the video will be assigned to the control group, so the study will be conducted over two groups. If the patient has watched the video; He will be asked whether he watches an animation video or a video with real surgery footage, and the reason for watching the video. Then, before starting the operation, they will be asked to score the sentences in the Situational and Trait Anxiety Inventory (Survey 2). By comparing the Situational Anxiety Inventory made at the time of the surgery appointment with the Situational Anxiety Inventory scores made just before the surgery. it will be evaluated whether the patients who watch videos have more anxiety. At the same time, it will be evaluated whether the patients who have a high Trait Anxiety Inventory score when making an appointment and who generally have high anxiety watch more videos. This study is planned to be performed on a total of 60 patients, 30 of whom watch videos and 30 who do not.

#### Survey 1

**Table 1: STAI-S Form (State Anxiety Test)** 

| | | None | A | A lot | Fully |
|---|---|---|---|---|---|
| | | | little | | - |
| one. | I am currently a resident. | (one) | (2) | (3) | (4) |
| 2. | I feel safe. | (one) | (2) | (3) | (4) |
| 3. | I'm nervous right now. | (one) | (2) | (3) | (4) |
| 4. | I feel regret. | (one) | (2) | (3) | (4) |
| 5. | I am at peace right now. | (one) | (2) | (3) | (4) |
| 6. | I'm not having any fun right now. | (one) | (2) | (3) | (4) |
| 7. | I worry about what will happen to me. | (one) | (2) | (3) | (4) |
| 8. | I feel rested. | (one) | (2) | (3) | (4) |
| 9. | I am anxious right now. | (one) | (2) | (3) | (4) |
| 10. | I feel comfortable. | (one) | (2) | (3) | (4) |
| 11th. | I have confidence. | (one) | (2) | (3) | (4) |
| 12. | I'm broke right now. | (one) | (2) | (3) | (4) |
| 13. | I'm so angry. | (one) | (2) | (3) | (4) |
| 14. | I feel my nerves are very tense. | (one) | (2) | (3) | (4) |
| 15. | I feel relieved. | (one) | (2) | (3) | (4) |
| 16. | I am content with my situation right now. | (one) | (2) | (3) | (4) |
| 17. | I am worried right now. | (one) | (2) | (3) | (4) |

**C.3** 

**C.2** 

| 18. | I feel stunned with excitement. | (one) | (2) | (3) | (4) |
|-----|---------------------------------|-------|-----|-----|-----|
| 19. | I am happy right now. | (one) | (2) | (3) | (4) |
| 20. | I'm in good spirits right now. | (one) | (2) | (3) | (4) |

Table 2: STAI-T Form (Trait Anxiety Test)

| | , | None | Α | A lot | Fully |
|---|---|---|---|---|---|
| | | | little | | - |
| 21. | I am usually in good spirits. | (one) | (2) | (3) | (4) |
| 22. | I usually get tired quickly. | (one) | (2) | (3) | (4) |
| 23. | I usually cry easily. | (one) | (2) | (3) | (4) |
| 24. | I want to be as happy as anyone else. | (one) | (2) | (3) | (4) |
| 25. | I miss opportunities because I can't decide quickly | (one) | (2) | (3) | (4) |
| 26. | I feel rested | (one) | (2) | (3) | (4) |
| 27. | usually calm, restrained and cool | (one) | (2) | (3) | (4) |
| 28. | I feel the difficulties pile up so much that I can't overcome | (one) | (2) | (3) | (4) |
| | them | | | | |
| 29. | I worry about unimportant things | (one) | (2) | (3) | (4) |
| 30. | I'm usually happy | (one) | (2) | (3) | (4) |
| 31. | I take everything seriously and worry | (one) | (2) | (3) | (4) |
| 32. | I'm usually insecure | (one) | (2) | (3) | (4) |
| 33. | I usually feel safe | (one) | (2) | (3) | (4) |
| 34. | I avoid facing difficult and difficult situations | (one) | (2) | (3) | (4) |
| 35. | I usually feel sad | (one) | (2) | (3) | (4) |
| 36. | I am generally satisfied with my life | (one) | (2) | (3) | (4) |
| 37. | Irrelevant thoughts bother me | (one) | (2) | (3) | (4) |
| 38. | I take disappointments so seriously that I can never forget | (one) | (2) | (3) | (4) |
| | them. | | | | |
| 39. | I am a sane and determined person | (one) | (2) | (3) | (4) |
| 40. | Things that have been on my mind lately are making me | (one) | (2) | (3) | (4) |
| | nervous. | | | | |

# Survey 2

| 1. | Have | you | watched | а | video | about | embedded | tooth | extraction | from | any | social | media |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| pla | atform | ? | | | | | | | | | | | |

□Yes □No

| 2. | Was the video v | you watched a real | l surgery vide | o or an | animation | video? |
|---|---|---|---|---|---|---|
| | TTUS LITE TIMES | you wateried a rea | i Juigoi y viuc | o oi aii | ammanom | VIGCO. |

□animation video

□Real surgery video

# 3. What is the reason for watching the video?

□To learn more about the operation.

☐ Preparing myself before the operation.

 $\hfill\square$  Because I'm afraid of the operation

□Other ( ...... )

# **STAI-S Form (Situational Anxiety Test)**

| | | None | A<br>little | A lot | Fully |
|------|----------------------------|-------|-------------|-------|-------|
| one. | I am currently a resident. | (one) | (2) | (3) | (4) |
| 2. | I feel safe. | (one) | (2) | (3) | (4) |

| 3. | I'm nervous right now. | (one) | (2) | (3) | (4) |
|-------|-------------------------------------------|-------|-----|-----|-----|
| 4. | I feel regret. | (one) | (2) | (3) | (4) |
| 5. | I am at peace right now. | (one) | (2) | (3) | (4) |
| 6. | I'm not having any fun right now. | (one) | (2) | (3) | (4) |
| 7. | I worry about what will happen to me. | (one) | (2) | (3) | (4) |
| 8. | I feel rested. | (one) | (2) | (3) | (4) |
| 9. | I am anxious right now . | (one) | (2) | (3) | (4) |
| 10. | I feel comfortable. | (one) | (2) | (3) | (4) |
| 11th. | I have confidence. | (one) | (2) | (3) | (4) |
| 12. | I'm broke right now. | (one) | (2) | (3) | (4) |
| 13. | I'm so angry. | (one) | (2) | (3) | (4) |
| 14. | I feel my nerves are very tense. | (one) | (2) | (3) | (4) |
| 15. | I feel relieved. | (one) | (2) | (3) | (4) |
| 16. | I am content with my situation right now. | (one) | (2) | (3) | (4) |
| 17. | I am worried right now. | (one) | (2) | (3) | (4) |
| 18. | I feel stunned with excitement. | (one) | (2) | (3) | (4) |
| 19. | I am happy right now. | (one) | (2) | (3) | (4) |
| 20. | I'm in good spirits right now. | (one) | (2) | (3) | (4) |

Table 2: STAI-T Form (Trait Anxiety Test)

| | | None | A<br>little | A lot | Fully |
|---|---|---|---|---|---|
| 21. | I am usually in good spirits. | (one) | (2) | (3) | (4) |
| 22. | I usually get tired quickly. | (one) | (2) | (3) | (4) |
| 23. | I usually cry easily. | (one) | (2) | (3) | (4) |
| 24. | I want to be as happy as anyone else. | (one) | (2) | (3) | (4) |
| 25. | I miss opportunities because I can't decide quickly | (one) | (2) | (3) | (4) |
| 26. | I feel rested | (one) | (2) | (3) | (4) |
| 27. | I am usually calm, restrained and cool | (one) | (2) | (3) | (4) |
| 28. | I feel the difficulties pile up so much that I can't overcome them | (one) | (2) | (3) | (4) |
| 29. | I worry about unimportant things | (one) | (2) | (3) | (4) |
| 30. | I'm usually happy | (one) | (2) | (3) | (4) |
| 31. | I take everything seriously and worry | (one) | (2) | (3) | (4) |
| 32. | I'm usually insecure | (one) | (2) | (3) | (4) |
| 33. | I usually feel safe | (one) | (2) | (3) | (4) |
| 34. | I avoid facing difficult and difficult situations | (one) | (2) | (3) | (4) |
| 35. | I usually feel sad | (one) | (2) | (3) | (4) |
| 36. | I am generally satisfied with my life | (one) | (2) | (3) | (4) |
| 37. | Irrelevant thoughts bother me | (one) | (2) | (3) | (4) |
| 38. | I take disappointments so seriously that I can never forget them. | (one) | (2) | (3) | (4) |
| 39. | I am a sane and determined person | (one) | (2) | (3) | (4) |
| 40. | Things that have been on my mind lately are making me nervous. | (one) | (2) | (3) | (4) |

# SUBJECT OF THE RESEARCH

C.3.1

(Check the appropriate box(s) below.)

| C.3.1.1 | Observational studies ( excluding observational drug studies and observational medical device studies ) | | | |
|---|---|---|---|---|
| C.3.1.2 | Survey studies ( survey ) | | | |
| C.3.1.3 | Retrospective archive scans such a | | | |
| C.3.1.4 | such as blood, urine, tissue, radiole | crobiology, pathology and radiology cogical image | | |
| C.3.1.5 | Research to be carried out with materials obtained during routine examination, examination, analysis and treatment processes | | | |
| C.3.1.6 | In vitro studies with cell and tissue | e cultures | | |
| C.3.1.7 | Studies to be carried out with genetic material for identification purposes other than gene therapy clinical studies | | | |
| C.3.1.8 | Research to be conducted within the | he boundaries of nursing activities | | |
| C.3.1.9 | Research on body physiology such | n as exercise | | |
| C.3.1.1<br>0 | Evaluation studies of living habits | | | $\boxtimes$ |
| C.3.1.1<br>1 | New scale development | | | |
| C.3.1.1<br>2 | If other, please specify ( eg neurol medical purpose): | ogical data for use in the social and hu | iman sciences (witho | ut a |
| | RESEARCH QUALITY | | | |
| C.3.2 | | Descriptive | | |
| | | cross-sectional | | |
| | | case-control | | |
| | Observational Studies | Prospective cohort | + | |
| | | retrospective cohort | | |
| | | Other (specify) | | |
| C.3.3 | | <b>TEER GROUP</b> (One of the critical peristics of the volunteer group. Please | | |
| C.3.3.1 | Estimated Number of Volunteers : | | | |
| C.3.3.2 | under 18 years old | | | |
| C.3.3.3 | over 18 years: | | | $\boxtimes$ |
| C.3.3.4 | Woman | | | $\boxtimes$ |
| C.3.3.5 | Male | | | $\boxtimes$ |
| C.3.3.6 | healthy volunteers | | | $\boxtimes$ |
| C.3.3.7 | patients | | | |
| C.3.3.8 | Disabled people | | | |

| C.3.3.9 | pregnant women | | | | | |
|---|---|---|---|---|---|---|
| C.3.3.1<br>0 | breastfe | eeding women | | | | |
| C.3.3.1<br>1 | emerge | ncy cases | | | | |
| C.3.3.1<br>2 | Student | ts | | | | |
| C.3.3.1<br>3 | seniors | | | | | |
| C.3.3.1<br>4 | If other | If other, please specify: | | | | |
| C.3.4 | RESEA | ARCH CENTER | | | | |
| | The res | earch will be carried out in Kütahya Health Sciences Universityry, Department of Oral, Dental and Maxillofacial Surgery. | y, Facult | y of | | |
| C.3.5 | <ul> <li>CRITERIA FOR INCLUSION</li> <li>Patients aged 18-45 years</li> <li>The patient does not have any systemic disease</li> <li>mesio-angular radiographic grade of impacted tooth according to Winter classification or 2 or 3 / B according to Pell and Gregory classification</li> </ul> | | | | | |
| <ul> <li>EXCLUSION CRITERIA</li> <li>Patients using antidepressants and anxiolytic drugs</li> <li>impacted tooth extraction/difficult tooth extraction</li> <li>Patients with systemic disease</li> <li>Female patients who are pregnant or breastfeeding</li> </ul> | | | | | | |
| C.3.6 | CONTROL GROUP (if any) Patients who did not watch the surgery video on any social media source before the impacted tooth extraction operation | | | | | |
| C.3.7 | PLACE OF SURVEY AND PERMISSION STATUS The research will be carried out in Kütahya Health Sciences University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery. The decision of the academic board and the approval of the Chief Physician were taken. | | | | | |
| C.3.8 | DATA COLLECTION TOOLS and FEATURES (if scales, questionnaires and other tools are intended to be used, Turkish validity, reliability and scoring methods should be written here.) Survey 1 Table 1: STAI-S Form (State Anxiety Test) | | | | | |
| | 25.5 | Law annually a maidant | | A<br>little | A lot | Fully |
| | one. | I am currently a resident. | | (2) | (3) | (4) |
| | 2.<br>3. | I feel safe. | | (2) | (3) | (4) |
| | ٥. | I'm nervous right now. | (one) | (2) | (3) | (4) |

| 4. | I feel regret. | (one) | (2) | (3) | (4) |
|---|---|---|---|---|---|
| 5. | I am at peace right now. | (one) | (2) | (3) | (4) |
| 6. | I'm not having any fun right now. | (one) | (2) | (3) | (4) |
| 7. | I worry about what will happen to me. | (one) | (2) | (3) | (4) |
| 8. | I feel rested. | (one) | (2) | (3) | (4) |
| 9. | I am anxious right now. | (one) | (2) | (3) | (4) |
| 10. | I feel comfortable. | (one) | (2) | (3) | (4) |
| 11th. | I have confidence. | (one) | (2) | (3) | (4) |
| 12. | I'm broke right now. | (one) | (2) | (3) | (4) |
| 13. | I'm so angry. | (one) | (2) | (3) | (4) |
| 14. | I feel my nerves are very tense. | (one) | (2) | (3) | (4) |
| 15. | I feel relieved. | (one) | (2) | (3) | (4) |
| 16. | I am content with my situation right now. | (one) | (2) | (3) | (4) |
| 17. | I am worried right now. | (one) | (2) | (3) | (4) |
| 18. | I feel stunned with excitement. | (one) | (2) | (3) | (4) |
| 19. | I am happy right now. | (one) | (2) | (3) | (4) |
| 20. | I'm in good spirits right now. | (one) | (2) | (3) | (4) |

**Table 2: STAI-T Form (Trait Anxiety Test)** 

| Table 2: | STAI-T Form (Trait Anxiety Test) | | | | |
|---|---|---|---|---|---|
| | | None | Α | A lot | Fully |
| | | | little | | |
| 21. | I am usually in good spirits. | (one) | (2) | (3) | (4) |
| 22. | I usually get tired quickly. | (one) | (2) | (3) | (4) |
| 23. | I usually cry easily. | (one) | (2) | (3) | (4) |
| 24. | I want to be as happy as anyone else. | (one) | (2) | (3) | (4) |
| 25. | I miss opportunities because I can't decide quickly | (one) | (2) | (3) | (4) |
| 26. | I feel rested | (one) | (2) | (3) | (4) |
| 27. | usually calm, restrained and cool | (one) | (2) | (3) | (4) |
| 28. | I feel the difficulties pile up so much that I can't overcome them | (one) | (2) | (3) | (4) |
| 29. | I worry about unimportant things | (one) | (2) | (3) | (4) |
| 30. | I'm usually happy | (one) | (2) | (3) | (4) |
| 31. | I take everything seriously and worry | (one) | (2) | (3) | (4) |
| 32. | I'm usually insecure | (one) | (2) | (3) | (4) |
| 33. | I usually feel safe | (one) | (2) | (3) | (4) |
| 34. | I avoid facing difficult and difficult situations | (one) | (2) | (3) | (4) |
| 35. | I usually feel sad | (one) | (2) | (3) | (4) |
| 36. | I am generally satisfied with my life | (one) | (2) | (3) | (4) |
| 37. | Irrelevant thoughts bother me | (one) | (2) | (3) | (4) |
| 38. | I take disappointments so seriously that I can never forget them. | (one) | (2) | (3) | (4) |
| 39. | I am a sane and determined person | (one) | (2) | (3) | (4) |
| 40. | Things that have been on my mind lately are making me nervous. | (one) | (2) | (3) | (4) |

| Survey 2 |
|---|
| 1. Have you watched a video about embedded tooth extraction from any social media platform? |
| □Yes □No |
| 2. Was the video you watched a real surgery video or an animation video? |
| □animation video |
| □Real surgery video |
| 3. What is the reason for watching the video? |
| ☐To learn more about the operation. |
| □ Preparing myself before the operation. |
| ☐ Because I'm afraid of the operation |

| Other | () | | | |
|---|---|---|---|---|
| | STAI-S Form (Situational Anxiety Test) | | | |
| | | None | A | A lot |
| | | TVOILE | little | Aiot |
| one. | I am currently a resident. | (one) | (2) | (3) |
| 2. | I feel safe. | (one) | (2) | (3) |
| 3. | I'm nervous right now. | (one) | (2) | (3) |
| 4. | I feel regret. | (one) | (2) | (3) |
| 5. | I am at peace right now. | (one) | (2) | (3) |
| 6. | I'm not having any fun right now. | (one) | (2) | (3) |
| 7. | I worry about what will happen to me. | (one) | (2) | (3) |
| 8. | I feel rested. | (one) | (2) | (3) |
| 9. | I am anxious right now. | (one) | (2) | (3) |
| 10. | I feel comfortable. | (one) | (2) | (3) |
| 11th. | I have confidence. | (one) | (2) | (3) |
| 12. | I'm broke right now. | (one) | (2) | (3) |
| 13. | I'm so angry. | (one) | (2) | (3) |
| 14. | I feel my nerves are very tense. | (one) | (2) | (3) |
| 15. | I feel relieved. | (one) | (2) | (3) |
| 16. | I am content with my situation right now. | (one) | (2) | (3) |
| 17. | I am worried right now. | (one) | (2) | (3) |
| 18. | I feel stunned with excitement. | (one) | (2) | (3) |
| 19. | I am happy right now. | (one) | (2) | (3) |
| 20. | I'm in good spirits right now. | (one) | (2) | (3) |
| | 2: STAI-T Form (Trait Anxiety Test) | | | |
| | | None | A | A lot |
| | | | little | |
| 21. | I am usually in good spirits. | (one) | (2) | (3) |
| 22. | I usually get tired quickly. | (one) | | (3) |
| 23. | I usually cry easily. | (one) | | (3) |
| 24. | I want to be as happy as anyone else. | (one) | | (3) |
| 25. | I miss opportunities because I can't decide quickly | (one) | | (3) |
| 26. | I feel rested | (one) | | (3) |
| 27. | usually calm, restrained and cool | (one) | | (3) |
| 28. | I feel the difficulties pile up so much that I can't overcome them | (one) | | (3) |
| 29. | I worry about unimportant things | (one) | | (3) |
| 30. | I'm usually happy | (one) | | (3) |
| 31. | I take everything seriously and worry | (one) | | (3) |
| 32. | I'm usually insecure | (one) | | (3) |
| 33. | I usually feel safe | (one) | | (3) |
| <i>33</i> . | I avoid facing difficult and difficult situations | (one) | | (3) |
| | ŭ | (one) | | (3) |
| 34. | I usually feel sad | | \_/_/ | |
| 34.<br>35. | I usually feel sad I am generally satisfied with my life | | (2) | (.5) |
| 34.<br>35.<br>36. | I am generally satisfied with my life | (one) | | (3) |
| 34.<br>35.<br>36.<br>37. | I am generally satisfied with my life Irrelevant thoughts bother me | (one) | (2) | (3) |
| 34.<br>35.<br>36. | I am generally satisfied with my life | (one) | (2) | |

PROCESSES AND VARIABLES TO BE USED IN THE RESEARCH (In this section, all the procedures you will follow in the research, data collection methods, dependent and independent variables will be written.)

C.3.9

| | STATISTICAL ANALYSIS METHOD (It will be done in SPSS, it is not a sufficient answer) |
|---|---|
| | The sample size of the study was determined by statistical power analysis (G Power Statistical Program), in which 60 people (at least 30 people for each group) should be reached with 95% confidence interval ±3 error margin. |
| C.3.10 | for Windows 22.00 statistical package program will be used to perform data analysis. Chi-square and Fisher's exact chi-square test will be used for descriptive statistics. The mean, standard deviation and frequency distribution of the data will be calculated as a percentage. |
| | Dependent and independent variables between the two groups will be analyzed by chi-square and Mann Whitney U tests . |
| | RESEARCH PERIOD |
| C.3.11 | <b>Research start date:</b> (01/09/2021) ( Please specify a fixed date from the ethics committee approval date) |
| | <b>Estimated duration of the research</b> (such as two and a half years, one year and three months): 1 year (01/09/2021-01/09/2022) |
| | RESOURCES |
| | *Full references of at least 3 sources related to the subject of the study must be specified below and must be provided in print in the application file. |
| C.3.12 | 1. Toledano-Serrabona, Jorge, et al. "Effect of an Informative Video on Anxiety and hemodynamics Parameters in Patients Requiring Mandibular Third Molar Extraction: A Randomized Clinical Trial." Journal of Oral and maxillofacial Surgery 78.11 (2020): 1933-1941. |
| | 2. Omezli, Mehmet Melih, Damla Torul, and Kadircan Kahveci. "does watching Videos increase the perioperative Anxiety in Patients Undergoing Third Molar surgery? A Randomized Trial." Journal of Oral and maxillofacial Surgery 78.2 (2020): 216-e1. |
| | 3.Kazancioglu, Hakki Oguz, et al. " does watching a video on third molar surgery increase patients 'anxiety level." Oral surgery, oral medicine, oral pathology and oral radiology 119.3 (2015): 272-277. |

# D. RESEARCH BUDGET\*\*\*

| RESEARCH EXPENSES: I | f NONE, put ⊠a cross in the box | |
|---|---|---|
| D.1 | Service from the research site: ( For example; ECG 3 times, CT 2 times) | NO |
| D.2 | Service procurement from outside the research site: ( For example; such as laboratory services) | NO |
| D.3 | to volunteers :<br>(such as transportation and light<br>lunch) | NO |
| D.4 | Other ( such as travel, surveyor, survey papers printing costs, consumables ): | NO |

| D.5 | Total budget of the research: | NO |
|---|---|---|
| | SOURCE OF RESEARCH BUDGET: NONE | |
| | University ( BAP ) Application Has Been Made. | |
| D.6 | training and research Hospital | |
| | The Scientific, Technical and Resear (TÜBİTAK) Application has been m | |
| | State Planning Organization (SPO) A | Application has been made. |
| | Company | |
| | Research team (Please tick the releva yourself) | ant box if it will be met by |
| | Other | |
| | SUPPORTING INSTITUTION / C | ORGANIZATION INFORMATION |
| | Name of Institution: | |
| D.3 | Address: | |
| | E-mail address: | |
| | Phone number: | |
| | Fax number: | |

<sup>\*\*\*\*</sup> Please do not leave blank, if not, indicate "no"

#### **COMMITMENT**

- That this project has not been presented to another ethics committee before as we presented it to your committee.
- The information in the application file is correct,
- The research will be carried out in accordance with the protocol, the relevant legislation, the Kütahya Health Sciences University Non-Interventional Ethics Committee Directive, the current Helsinki Declaration and Good Clinical Practices.
- In the event that the research is not started or the research is abandoned within 6 (six) months from the date of approval by the Ethics Committee, we will inform your committee about the subject.
- of changes in the research team and changes in the research protocol, such as the purpose, method, etc., before the said change is made.
- we will submit the "research result report" and a full-text copy of the article when it is published to the Non-Interventional Ethics Committee of Kütahya Health Sciences University.
- We undertake that no non-routine transaction costs such as tests, laboratory examinations, physician examinations, use of chemicals and medical devices, etc. to be carried out within the scope of the research, will be covered or made to be paid by the public funds and budgets or private health insurances, and that the said costs will be paid by the person or organization supporting the project.

The section below will be filled in by handwriting.

The ranking below is not binding on the Author ranking at the time of publication.

Date:... / .... / 20

1. Name and surname: 6. Name and surname:

| | Signature: | | Signature : |
|----|------------------------------|-----|------------------------------|
| 2. | Name and surname: Signature: | 7. | Name and surname: Signature: |
| 3. | Name and surname: Signature: | 8. | Name and surname: Signature: |
| 4. | Name and surname: Signature: | 9. | Name and surname: Signature: |
| 5. | Name and surname: Signature: | 10. | Name and surname: Signature: |

# résumés

It belongs to all researchers participating in the study.

### 1. PERSONAL INFORMATION

| NAME, SURNAME: Dr. Instructor Member<br>Berkan ALTAY | DATE and PLACE OF BIRTH: 16.09.1991-Ankara |
|---|---|
| CURRENT POSITION: Dr. Faculty Member CORRESPONDING ADDRESS: Kütahya Universi and Research Center Directorate Faculty, Departme Lala Hüseyin Paşa Caddesi No:271 PK 43100 KÜT | ty of Health Sciences Oral and Dental Health Application nt of Oral and Maxillofacial Surgery, İstiklal Mahallesi AHYA |
| PHONE: 05356557441 E-MAIL: berkan.altay@ksbu.edu.tr | |

# 2. EDUCATION

| DEGREE | UNIVERSITY | FIELD OF LEARNING |
|---|---|---|
| Bachelor/Master | Kırkkale University<br>Faculty of Dentistry | Clinical Sciences |
| Expertise | Kırkkale University<br>Faculty of Dentistry | Oral, Dental and Maxillofacial Surgery |

#### 3. ACADEMIC EXPERIENCE

| TITLE | SECTION | UNIVERSITY |
|---|---|---|
| Research Assistant | Oral, Dental and<br>Maxillofacial Surgery | Kırkkale University Faculty of Dentistry (2016-2020) |
| Dr. Faculty Member | Oral, Dental and<br>Maxillofacial Surgery | Küyahya University of Health Sciences (2020-) |

#### 4. WORKING AREAS

| WORKING AREA | KEY WORDS |
|---|---|
| Oral, Dental and Maxillofacial Surgery | Implant surgery, oral surgery, bone healing, Maxillofacial trauma, TMJ surgery, Orthognathic surgery |

#### 5. IMPORTANT PUBLICATIONS IN THE LAST FIVE YEARS

- 1-Altay B, Dede EÇ, Ozgul O, Atıl F, Kocyigit ID, Orhan K, Tekin U, Korkusuz P, Önder ME, Effect of Systemic Oxytocin Administration on New Bone Formation and Distraction Rate in Rabbit Mandible, Journal of Oral and Maxillofacial Surgery (2020), doi: https://doi.org/10.1016/j.joms.2020.03.005.
- 2-Ozkan Ozgul , Berkan Altay, Fethi Atil , M. Ercument Leader , Hope Tekin , Seda Yilmaz , and Ismail Doruk cocyigit . Allogenic versus Autogenous Bone Rings in Dental Implant Surgery: Guidance of Stress Analysis-Part II. Journal of Biomaterials and Tissue Engineering Vol. 8, 448–453, 2018
- 3- Sanli E, Altay B. Pediatric dog bite injuries of head and neck: An algorithm for the treatment of our clinic. Turk J Plast Surg 2020; 28:51-4.

#### 6. PUBLICATIONS RELATED TO THE RESEARCH SUBJECT

#### 1. PERSONAL INFORMATION

| NAME, SURNAME: Dr. Instructor Member<br>Mohammad Nabi BASIRY | DATE and PLACE OF BIRTH: 27.06.1981 Kabul |
|---|---|
| CURRENT POSITION: Dr. Faculty Member | |
| CORRESPONDING ADDRESS: Kütahya University of Health Sciences Oral and Dental Health Application | |

CORRESPONDING ADDRESS: Kütahya University of Health Sciences Oral and Dental Health Application and Research Center Directorate Faculty, Department of Oral and Maxillofacial Surgery, İstiklal Mahallesi Lala Hüseyin Paşa Caddesi No:271 PK 43100 KÜTAHYA

PHONE: 05079321384

E-MAIL: mohammednabi.basiry@ksbu.edu.tr

#### 2. EDUCATION

| DEGREE | UNIVERSITY | FIELD OF LEARNING |
|---|---|---|
| Doctorate | Gulhane Military<br>Medical Academy | Oral, Dental and Maxillofacial Surgery |
| Degree | Kabul Medical<br>University / Faculty of<br>Stomatology (Dentistry) | Dentist |

#### 3. ACADEMIC EXPERIENCE

| TITLE | SECTION | UNIVERSITY |
|---|---|---|
| Dr. Instructor Member of | Oral, Dental and<br>Maxillofacial Surgery | Kütahya University of Health Sciences |
| Faculty Member | Oral, Dental and<br>Maxillofacial Surgery | Küyahya University of Health Sciences |

#### 4. WORKING AREAS

| WORKING AREA | KEY WORDS |
|---|---|
| Oral, Dental and Maxillofacial Surgery | Oral cancers, Oral diseases, Maxillofacial traumatology |
| | Oral Implantology |

#### 5. IMPORTANT PUBLICATIONS IN THE LAST FIVE YEARS

#### 6. PUBLICATIONS RELATED TO THE RESEARCH SUBJECT

#### 1. PERSONAL INFORMATION

| NAME, SURNAME: Dt . Shayma KALE | DATE and PLACE OF BIRTH: 22.03.1995-Kütahya |
|---|---|

CURRENT POSITION: Research Assistant

CORRESPONDENCE ADDRESS: Kütahya University of Health Sciences Oral and Dental Health Application and Research Center Directorate Faculty, Department of Oral and Maxillofacial Surgery, İstiklal Mahallesi Lalahüseyinpaşa Caddesi No:271 PK 43100 KÜTAHYA

PHONE: 05533618111

E-MAIL: seyma.kale@ksbu.edu.tr

#### 2. EDUCATION

| DEGREE | UNIVERSITY | FIELD OF LEARNING |
|--------|------------|-------------------|
|--------|------------|-------------------|

| Licence | Eskişehir Osmangazi<br>University Faculty of<br>Dentistry | Dentist |
|---|---|---|
| | • | |

#### 3. ACADEMIC EXPERIENCE

| TITLE | SECTION | UNIVERSITY |
|---|---|---|
| Research Assistant | Dentistry-Oral and<br>Maxillofacial Surgery | Kütahya University of Health Sciences |

#### 4. WORKING AREAS

| WORKING AREA | KEY WORDS |
|---|---|
| Oral, Dental and Maxillofacial Surgery | Oral anatomy, oral cancers, dental implant |

#### 5. IMPORTANT PUBLICATIONS IN THE LAST FIVE YEARS

#### 6. PUBLICATIONS RELATED TO THE RESEARCH SUBJECT

# FOR "NON-INTERVENTIONAL CLINICAL TRIALS" INFORMED VOLUNTARY CONSENT FORM

**Name of the Research Project:** Evaluation of the Effect of Watching Videos on Social Media on Anxiety Before Impacted Wisdom Tooth Extraction

Name of Responsible Investigator: Dr. Instructor Member Berkan Altay Name of Other Researchers: Dr. Mohammad Nabi Basiry , Dt . Seyma Castle

**Supporter (if applicable):** 

You have been invited to take part in a study titled "The Evaluation of the Effects of Watching Videos on Social Media on Anxiety Before Impacted Wisdom Tooth Extraction". The aim of this study is to evaluate the effects of watching videos with surgical images on social media on anxiety before the impacted tooth extraction operation. This study is conducted for research purposes and participation is on a voluntary basis. We would like to inform you about the research before you decide to participate in the study. Once you are fully informed about the study and your questions have been answered, you will be asked to sign this form if you wish to participate. This research was carried out in the Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery, Dr. It is under the responsibility of Faculty Member Berkan Altay.

What is the purpose of the study; How many people other than me will participate in this study? The following information should be included under this heading:

- social media before the impacted tooth extraction operation on anxiety,
- 60 people who applied to our hospital and volunteered to participate in the study.

#### Should I participate in this study? (This section will be preserved as it is)

Whether or not you participate in this study is entirely up to you. Even if you sign this form now, you are free to stop working at any time without giving a reason. If you do not want to participate or leave the study, the most appropriate treatment plan for you will be applied by your doctor. Likewise, the doctor conducting the study may decide that it will not be beneficial for you to continue the study and may exclude you from the study, in which case the most appropriate treatment will be chosen for you.

#### What awaits me if I participate in this study?

If you participate in this study, you will be asked to fill out two questionnaires in total, at the session we made an appointment for impacted tooth extraction and just before the surgery. The surveys will be made only once and will not need to be repeated.

#### Are there risks and inconveniences to the work?

No interventional procedure will be required in our study. For this reason, you will not feel any risk and discomfort.

#### What are the benefits of taking part in the study?

As a result of the research, it will be determined whether watching surgery videos on social media before impacted tooth extraction surgery is effective on anxiety and if so, in what way.

#### What is the cost of participating in this study? (This section will be preserved as it is)

You will not be under any financial burden by participating in the study and you will not be paid any money.

#### How will my personal information be used? (This section will be preserved as it is)

Your study doctor will use your personal information to conduct the research and statistical analysis, but your identity will be kept confidential. Ethics committees or official authorities may review the information about you only if necessary. At the end of the study, you have the right to ask for information about your own results. Study results will be published in the medical literature at the end of the study, but your identity will not be disclosed.

#### Who can I contact for more information?

If you need additional information about the study, please contact the person below.

NAME: Dr. Berkan Altay

POSITION: Dr. Faculty Member MOBILE PHONE: +90(535)655 7441

NAME: Dr. Mohammad Nabi Basiry

**POSITION: Dr. Lecturer** 

MOBILE PHONE: +90(507)932 1384

NAME: Dt. Shayma KALE POSITION: Research Assistant MOBILE PHONE: +90(553)3618111

#### (Participant/Patient Statement)

Dr. Faculty Member Berkan ALtay stated that a medical research would be conducted in the Department of Oral, Dental and Maxillofacial Surgery, Faculty of Dentistry, Kütahya Health Sciences University, and the above information about this research was conveyed to me and I read the relevant text. After this information, I was invited to such a research as a "participant". I have not encountered any compelling behavior regarding my participation in the research. I also know that if I refuse to participate, it will not do any harm to my medical care and my relationship with my physician. During the execution of the project, I can withdraw from the research without giving any reason. (However, I am aware that it would be appropriate to inform the researchers in advance that I would withdraw from the research in order not to put the researchers in a difficult situation). I may also be

excluded from the research by the researcher, provided that no harm is done to my medical condition. I do not take any financial responsibility for the expenses to be made for the research. I will not be paid either. I understand that the confidentiality of personal information about me obtained from the research will be protected. Necessary assurance was given that in case of any health problems that may arise due to the research practice, all kinds of medical interventions will be provided. (I will not be financially burdened with these medical interventions either). When I encounter a health problem during the research; at any hour, Dr.Berkan ALTAY +90(535)655 74, Dr. Mohammad Nabi Basiry +90(507)932 1384, Dt.Şeyma KALE +90(553)361 81 11(Kütahya Health Sciences I know that I can call from İstiklal Mahallesi Lalahüseyinpaşa Caddesi No:271 43100 KÜTAHYA), Department of Oral and Maxillofacial Surgery, Directorate of Oral and Dental Health Application and Research Center of the University. (Doctor's name, telephone and address information must be specified)

I have fully understood all the explanations given to me. I hereby agree to participate voluntarily in the clinical trial in question, of my own free will, without any pressure or coercion.

A copy of this signed form paper will be given to me.

| P | ar | ti | ci | n | ล | n | t |
|---|----|----|----|---|---|----|---|
| • | aı | u | L | μ | а | 11 | ı |

Name and surname:

Address: Phone: Signature: History:

#### interview witness

Name and surname:

Address: Phone: Signature: History:

#### Participant with interviewing physician

Name, surname, title:

Address: Phone: Signature: History:

LIGHTING AND THE STATEMENT OF THE PARTICIPANT WILL DEFINITELY BE THE CONTINUATION OF EACH OTHER. IT WILL NOT BE AVAILABLE ON SEPARATE PAGES.

| GOOD CLINICAL PRACTICE, GOOD LABORATORY PRACTICE AND HELSINKI<br>DECLARATION |
|---|
| COMMITMENTS |
| History |
| Name of the Study: Evaluation of the Effect of Watching Videos on Social Media on Anxiety Before Impacted Wisdom Tooth Extraction |
| TR Health by the Ministry; into effect Good Clinic _ Practices (ICU) and Good Laboratory Applications (ILU) Guides with the Declaration of Helsinki last published version I read . Above First Name last study This your guides to the principles suitable will do commitment I will . |
| Responsible Researcher : Dr. Berkan ALTAY Signed : |

Helper Researcher (s) : Dr. Mohammad Nabi BASIRY Signature :

Dt. Şeyma KALE Signature :